CLINICAL TRIAL: NCT02524834
Title: Proposed Single Center Investigational Device Exemption: Endovascular Repair of Descending ThoracoAbdominal Aortic Pathologies Using Physician Modified Endovascular Prosthesis
Brief Title: Endovascular Repair of Descending ThoracoAbdominal Aortic Pathologies Using Physician Modified Endovascular Prosthesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: Rodney A. White, MD (Other)
Collaborators: Long Beach Memorial Medical Center (Other)
Responsible Party: Sponsor-Investigator, Rodney A. White, MD, Medical Director, Vascular Surgery, Long Beach Memorial Heart & Vascular Institute, Long Beach, CA, MemorialCare Health System
Organization: MemorialCare Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSIDE:Thoracoabdominal Lesions
Record Dates: First submitted 2015-07-31; First posted 2015-08-17 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Aortic Disease
Keywords: Thoracoabdominal lesions
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Endovascular Device Implantation (Experimental): Endoluminal exclusion of thoracoabdominal lesion
  Interventions: Procedure: Exclusion of thoracoabdominal lesion; Device: Endovascular Device Implant

INTERVENTIONS:
Procedure: Exclusion of thoracoabdominal lesion — Endovascular repair of thoracoabdominal lesion with a physician modified Medtronic Valiant stent graft
Device: Endovascular Device Implant — Endovascular repair of thoracoabdominal lesion with a physician modified Medtronic Valiant stent graft

SUMMARY:
This is an early feasibility study that investigates the outcome of selected patients with complex thoracoabdominal aortic lesions who are suitable for endovascular (within the vessel) repair with a physician-modified Medtronic Thoracic Valiant stent graft. The Medtronic Valiant System includes a Valiant Thoracic Stent Graft, a self-expanding, tubular end prosthesis which is modified/customized by the Investigators to fit the patient's anatomy. The device is constructed by making a taper in the larger proximal thoracic device and attaching it to a smaller distal thoracic device. The Viabahn branches for the visceral vessels are sutured to holes made in the tapered section. The modified Valiant stent graft is advanced to the lesion site endoluminally via the iliac/femoral artery. Access for delivery of extensions to the device will be delivered through the left subclavian artery. Upon deployment, the stent graft self-expands at the target location, where it is designed to exclude the lesion by restoring blood flow through the stent graft lumen.

DETAILED DESCRIPTION:
The study will be conducted with non-surgical or very high-risk patients who are considered suitable candidates for endoluminal repair and who are diagnosed with a Type IV complex thoracoabdominal aortic lesion. The total number of enrolled subjects is planned to be 15. It is a prospective evaluation of patients receiving the device to determine the proportion in whom successful implantation is achieved, as indicated by exclusion of the thoracic lesion and graft patency at implant, time of discharge, and 1, 6, and 12 months following implantation, and to determine the proportion of patients who die or experience adverse events during and after the implantation. Furthermore, the percentage of patients in whom technical and clinical success is achieved, will be determined. Patients will be followed for 5 years after the surgery in which the stent graft is implanted.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Type IV complex thoracoabdominal aortic lesion and be considered candidates for endovascular repair;
* Patients must have an ileofemoral access compatible with delivery of a 25 Fr MedtronicValiant thoracic endograft;
* Patients must have a left subclavian artery anatomy compatible with 8 mm Dacron conduit to provide safe, sequential antegrade deployments of branch extensions
* Patients must have a nonaneurysmal proximal aortic segment distal to the left subclavian artery with at least 2 cm length to assure secure proximal fixation with a

  * Minimum diameter of 28 mm
  * Maximum diameter of 42mm
  * Angle less than 60° relative to axis of the aneurysm
  * Angle less than 60° relative to axis of the thoracic aorta;
* Patients must have a distal fixation iliac artery diameter greater than 2 cm in length and 12-28 mm in diameter;
* Patients must be high-risk surgical candidates according to the following established criteria: ASA score of IV.

Exclusion Criteria:

* Pregnant or pediatric patients (younger than 21 years of age);
* Patients who have a condition that threatens to infect the stent graft/aortic valve prosthesis;
* Patients with allergies to the stent graft material;
* Patients who fail to sign informed consent;
* Patients with expected survival less than one year.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days post intervention
  Early (at 30-days) death
Additional endovascular procedure | At 30 days
  Re-intervention
Conversion to open repair | At 30 days
  Surgical conversion
Stroke | At 30 days
  Stroke
All cause mortality | At 1 year post procedure
  Death
Additional endovascular procedure | At 1 year
  Re-intervention
Conversion to open repair | At 1 year
  Surgical conversion

SECONDARY OUTCOMES:
Vessel complications | Up to 5 years post intervention
  Includes dissection, thrombosis, embolization of vessels, malperfusion of branch vessels
Technical observations | Up to 5 years post intervention
  Includes loss of patency, endoleaks, twisting, kinking, fracture of stent graft, migration and separation of components
Composite of myocardial infarction, organ failure, sepsis | Up tp 5 years post intervention
  Includes Myocardial Infarction, organ failure and sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A White, MD, Principal Investigator — Medical Director, Vascular Surgery Long Beach Memorial Heart & Vascular Institute, Long Beach, CA
Locations (1):
- Long Beach Memorial Medical Center, Memorial Heart & Vascular Institute, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No